CLINICAL TRIAL: NCT05767450
Title: Assessing the Role of the Gut Microbiome and of the Intestinal Barrier Integrity in the Immune Pathogenesis of Type 1 Diabetes
Brief Title: Intervention on New Onset-T1D Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marika Falcone, Group Leader, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2019-123-70721
Record Dates: First submitted 2022-11-21; First posted 2023-03-14 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes
Keywords: Gut microbiome; Intestinal barrier integrity
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Interventional, randomized (1:1), 2-arm, single-center, placebo controlled
Who Masked: Participant
Masking Description: Participants will be randomized in blind (by a computer) in 1:1 allocations. Participants enrolled in both arms and their parents wil be blinded to treatment as sachets provided will be identical as will be the visual aspect and taste of the Vivomixx probiotic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated (Experimental): Probiotic name: Vivomixx® Form: powder Dosage: 4,4g/sachet with 450 billion of lactobacilli and bifidobacteria in a base of maltose Frequency: 1 sachet/day for children <10 year old or 2 sachets/day for children >10 year old Duration: 90 days
  Interventions: Dietary Supplement: Probiotic Vivomixx®
- Untreated (Placebo Comparator): Product name: Placebo Form: powder Dosage: 4,4g/sachet containing maltose Frequency: 1 sachet/day for children <10 year old or 2 sachets/day for children >10 year old Duration: 90 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Vivomixx® — The correct number of Vivomixx® sachets are given to parents with the indication to administer the dietary supplement as dissolved in drinking water or non-carbonated drinks.
  Other Names: VSL#3; Visbiome®
  Arms: Treated
Dietary Supplement: Placebo — The correct number of Placebo sachets are given to parents with the indication to administer the dietary supplement as dissolved in drinking water or non-carbonated drinks.
  Arms: Untreated

SUMMARY:
A pilot proof of concept clinical trial will be performed to demonstrate the restoration of gut barrier integrity by administration of beneficial anti-inflammatory gut microbial strains (Lactobacilli-enriched Vivomixx® probiotic) to new onset Type 1 Diabetes Children.

DETAILED DESCRIPTION:
This is an interventional randomized, 2-arm, single-blind, single-center, placebo-controlled mechanistic clinical trial (1:1).

One sachet of probiotic for children < 10 years old or two sachets for subjects > 10 years old dissolved into water or noncarbonated drinks will be administered every day for 90 consecutive days.The primary end point of the study will be the preservation of the residual insulin-producing beta-cell mass measured as the change in C-peptide values at 12 months after the beginning of treatment. Moreover, the investigators will collect blood samples for serological analysis (autoantibodies detection, measurement of biomarkers of gut barrier integrity) and immunological profiling; fecal samples for microbiome and metabolomic analysis. Finally the investigators will assess whether the response to Vivomixx® probiotic remains stable over a long-term period, that is in the absence of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of insulin-dependent type 1 diabetes
* Positive for at least one islet autoantibody (ICA, GADA, IA-2, IAA, ZnT8)
* No more than 3 months from first insulin injection
* ≥ 7 to < 18 year old

Exclusion Criteria:

* Diagnosed with celiac disease, IBD or other intestinal inflammatory pathologies
* Diagnosed with tuberculosis, hepatitis B or C, HIV, or active EBV or CMV infection; significant cardiac disease; conditions associated with immune dysfunction or hematologic dyscrasia (including malignancy, lymphopenia, thrombocytopenia, or anemia); liver or renal dysfunction.
* Ongoing use of systemic medications other than insulin.
* Recent administration of antibiotics (1 months prior to treatment)
* Deemed unlikely or unable to comply with the protocol or have any complicating medical issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Preservation of the residual insulin-producing beta cell mass | through study completion, an average of 1 year
  The primary outcome of the study will be the preservation of the residual insulin-producing beta-cell mass in newly diagnosed T1D patients that received the probiotic Vivomixx® in comparison to those receiving placebo. This parameter will be reported as the change in C-peptide values (ng/mL) before starting treatment (baseline) and 12 months after treatment initiation.
Glycemic control by Time-in-Range (TIR) monitoring | through study completion, an average of 1 year
  Glycemic control will be monitored in newly diagnosed T1D patients that received the probiotic Vivomixx® in comparison to those receiving placebo. This parameter will be reported as the change in TIR values (%) - that is the percentage of time in which blood glucose (blood sugar) remains in the safe target range of 70-180mg/dL - recorded before starting treatment (baseline) and 12 months after treatment initiation.

SECONDARY OUTCOMES:
Gut barrier integrity | through study completion, an average of 1 year
  The levels of zonulin and LBP will be measured in the serum before starting Vivomixx® or placebo administration (baseline), 3 months and 6 months after treatment initiation, as biomarkers used to determine the integrity of the intestinal epithelium in humans.
Gut microbiome profile | through study completion, an average of 1 year
  The gut microbiota composition will be analyzed on fecal samples collected before starting Vivomixx or placebo administration (baseline), 3 months and 6 months after treatment, 16S ribosomal RNA (rRNA) sequencing.
Measurement by flow cytometry of differences in the percentages of regulatory and inflammatory CD4 T cells | through study completion, an average of 1 year
  Changes in circulating regulatory and inflammatory CD4 T cell subsets (Treg, Th1, Th2, Th17) will be evaluated by flow cytometry of the expression of:
  * CD4, FOXP3 (Treg)
  * CD4, CRTH2 (Th2)
  * CD4, Tbet (Th1)
  * CD4, RORgt (Th17)
  Results will be expressed in term of percentage (%) of CD4 T cells expressing the molecules
Measurement by flow cytometry of differences in the percentages of MAIT cells and TCR gamma Delta T cells | through study completion, an average of 1 year
  Changes in circulating MAIT and TCR gammaDelta T cell subsets will be evaluated by flow cytometry of the expression of CD3, TCRgD, CD161, TCRva7.2
  Results will be expressed in term of percentage (%) of cells expressing CD3, TCRgD molecules (that are TCRgammaDelta T cells) and CD3, CD161, TCRva7.2 molecules (that are MAIT cells)
Measurement by flow cytometry of differences in the percentages of innate lymphoid cells | through study completion, an average of 1 year
  Changes in circulating MAIT and TCR gammaDelta T cell subsets will be evaluated by flow cytometry of the expression of Lineage markers, c-kit, CRTH2
  Results will be expressed in term of percentage (%) of Lineage-negative cells expressing c-kit or CRTH2 molecules.

CONTACTS AND LOCATIONS:
Overall Officials: Marika Falcone, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Autoimmune Pathogenesis Unit, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolpady J, Sorini C, Di Pietro C, Cosorich I, Ferrarese R, Saita D, Clementi M, Canducci F, Falcone M. Oral Probiotic VSL#3 Prevents Autoimmune Diabetes by Modulating Microbiota and Promoting Indoleamine 2,3-Dioxygenase-Enriched Tolerogenic Intestinal Environment. J Diabetes Res. 2016;2016:7569431. doi: 10.1155/2016/7569431. Epub 2015 Dec 8. PMID 26779542
- [Background] Caballero-Franco C, Keller K, De Simone C, Chadee K. The VSL#3 probiotic formula induces mucin gene expression and secretion in colonic epithelial cells. Am J Physiol Gastrointest Liver Physiol. 2007 Jan;292(1):G315-22. doi: 10.1152/ajpgi.00265.2006. Epub 2006 Sep 14. PMID 16973917
- [Background] Korpela R, Niittynen L. Probiotics and irritable bowel syndrome. Microb Ecol Health Dis. 2012 Jun 18;23. doi: 10.3402/mehd.v23i0.18573. eCollection 2012. PMID 23990830